CLINICAL TRIAL: NCT06861127
Title: Role of MRI in Diagnosis of Postpartum Neurological Disorders
Status: Active, not recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Petet Gadallah Nazir, Peter Gadallah, Sohag University
Other Study IDs: Soh-Med--25-1-01MS
Record Dates: First submitted 2025-02-18; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-09

CONDITIONS: Role of MRI in Diagnosis of Postpartum Neurological Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Role of MRI in diagnosis of postpartum neurological disorders

ELIGIBILITY:
Inclusion Criteria:

1. Female gender.
2. Age more than 18 years old.
3. Patients presented with neurological complaint in 3 months following childbirth.

Exclusion Criteria:

1. Male gender.
2. Female younger than 18 years old
3. Contraindication to perform MRI examination. These include:- Cardiac pacemaker.- Metallic aneurysm clips.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: 50
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-10-02 (Estimated); Study Completion 2025-10-02 (Estimated)

PRIMARY OUTCOMES:
Distribution of MRI Abnormalities in Postpartum Neurological Cases | 16 months
  This outcome measures the number of postpartum patients presenting with different types of MRI abnormalities, including PRES (Posterior Reversible Encephalopathy Syndrome), cerebral venous thrombosis, and other neurological conditions. The study aims to categorize and quantify these findings to better understand their prevalence and role in postpartum neurological disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Sohag Governorate, Egypt